CLINICAL TRIAL: NCT00707486
Title: A Randomized, Self Controlled Clinical Study of Hemostatic Efficacy of the HemCon Dental Dressing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2007-I-D-1
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-12

CONDITIONS: Tooth Extractions
Keywords: Hemostasis, tooth extractions, third molar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemcon Dental Dressing (Experimental): The HemCon® Bandage is an FDA-cleared chitosan-based flat bandage that controls severe arterial bleeding from traumatic injuries. In comparison to traditional bandages, the HemCon® Bandage provides superior control of bleeding, wound site adhesiveness, multiple injury site usage, biocompatibility and provides a barrier to infective agents.
  Interventions: Device: Hemcon Dental Dressing
- Gauze with pressure and/or Gelfoam (Active Comparator): Post operative care for oral surgery subjects consists of the subject biting on sterile cotton gauze to provide pressure to the extraction site. A common alternative practice involves the placement of Gelfoam (with or without antibiotic/steroid medication) into the extraction socket prior to application of the sterile gauze pressure dressing. This treatment was chosen as the study control to compare the HemCon Dental Dressing to the standard of care for oral surgery subjects, including the use of cotton gauze and/or Gelfoam to control post operative bleeding.
  Interventions: Device: Gauze with Pressure and/or Gelfoam

INTERVENTIONS:
Device: Hemcon Dental Dressing — The Hemcon Dental Dressing is an oral wound dressing made of chitosan.
  Arms: Hemcon Dental Dressing
Device: Gauze with Pressure and/or Gelfoam — Common practice for oral surgery patients involves the use of sterile dressing over the extraction site. The subject will provide the pressure by biting down on the sterile gauze. As previously discussed, other practices involve the use of Gelfoam prior to application of sterile gauze.
  Arms: Gauze with pressure and/or Gelfoam

SUMMARY:
The purpose of this study is to determine if the HemCon Dental Dressing is effective in stopping bleeding during dental surgeries.

DETAILED DESCRIPTION:
The HemCon® Bandage has been successfully used to achieve hemostasis in patients with high systolic pressure, high blood volume wounds, and to promote hemostasis on a massive scale compared to the hemostasis requirements of oral surgery wounds. Therefore, a human clinical trial has recently been completed evaluating the efficacy of using the HemCon® Bandage in a smaller finished size for dental extraction and other oral surgery sites. The HemCon® Bandage was proven to be significantly better at promoting hemostasis of oral surgery wounds than the control (cotton gauze or Gelfoam) in all subjects tested. All HemCon® Bandage sites achieved hemostasis faster than the control sites. Based on this data, a 510(k) was submitted and has received FDA clearance for the HemCon® Dental Dressing to be used as an oral wound dressing intended as a physical barrier for temporary protection of oral mucosal tissue and to provide pain relief.

This study evaluates the FDA cleared HemCon® Dental Dressing for use in hemostasis of soft oral tissue subsequent to dental surgical procedures such as tooth extractions excluding procedures involving primary closure of the HemCon® Dental Dressing within the oral wound.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring 2 or 4 3rd molar tooth extraction procedures.
* Index pairing must reflect anatomically similar extraction locations, i.e., for 2 extractions both must be upper or both must be lower extractions.
* Patients must be 14 years of age or older
* Patients must be available for a minimum of one post operative evaluation to be scheduled at the time of the procedure approximately 7 days post surgery. Additional follow-up visits may be scheduled at the discretion of the surgeon based on the severity of particular patient cases or the patient's need for earlier follow-up.
* Extraction sites do not require primary closure or suturing
* Willingness and ability to provide informed consent/ assent for participation
* Patients with seafood allergies
* Patients who have discontinued the use of anticoagulant medications (e.g., aspirin, coumadin, Plavix, etc.) for a minimum of 3 days prior to their planned surgical visit.

Exclusion Criteria:

* Scheduled to undergo a surgical procedure other than 3rd molar tooth extractions
* Scheduled to undergo 2 extractions whereby one is an upper 3rd molar and the other is a lower 3rd molar. These will not reflect a proper index pairing for statistical calculations and data analysis based on anatomical similarities.
* Extraction procedures are expected to require primary closure or suturing of the HemCon® Dental Dressing within the oral wound.
* Unable or unwilling to provide informed consent/ assent for participation as a subject
* Patients who are currently taking anticoagulant medications (e.g., aspirin, coumadin, Plavix, etc.) or have discontinued their anticoagulant medications less than 3 days prior to their surgical visit.
* Patients who are undergoing bisphosphonate therapy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay P Malmquist, DMD, Principal Investigator
Locations (2):
- United States (2):
  - Rodney Nichols, DMD, Milwaukie, Oregon
  - Jay P. Malmquist, DMD, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited as they presented at the site of the study for extraction. Subjects served as their own control as they had four extractions per procedure and two served as the experimental sites and two served as the control sites.
Groups:
- Hemcon Dental Dressing With Pressure: Subjects served as their own control. Subject had both the HemCon Dental Dressing and one of two controls: Gelfoam or Gauze with pressure. Subjects had paired extractions; each extraction site within the pair were randomized to the HemCon Dental Dressing or to a control.
Period: Overall Study
Arm/Group | Hemcon Dental Dressing With Pressure
Started | 72
Completed | 71
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Hemcon Dental Dressing and Gauze With Pressure: In the case of this study, participants served as their own control.
Arm/Group | Hemcon Dental Dressing and Gauze With Pressure
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 42
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 19.1 (3.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 72
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73.3 (8.36)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 128.1 (15.13)

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: This outcome measures the time it takes in minutes for the subject's extraction site to stop bleeding. It is divided by intervention.
Time Frame: Minutes After Application
Population: Participants served as their own control thus the total amount of participants is reflected in both of the outcome measures.
Measure: Mean (Standard Error); unit: Minutes
Units Other Than Participants: Extraction Sites
Groups:
- HemCon: Experimental
Arm/Group | HemCon | Control: Gauze | Total
Number analyzed (Participants) | 71 | 71 | 71
Number analyzed (Extraction Sites) | 140 | 140 | 280
Minutes | 1.9 (1.36) | 9.8 (3.96) | 6.0 (5.09)

2. Secondary Outcome: Incidence of Post Surgical Sequelae
Time Frame: 1 week post surgery
Measure: Number; unit: Percent of Participants
Arm/Group | HemCon | Control: Gauze | Total
Number analyzed (Participants) | 34 | 18 | 68
Percent of Participants
  Pain Score: None | 41.2 | 55.6 | 41.2
  Pain Score: Mild | 38.2 | 38.9 | 44.1
  Pain Score: Moderate | 14.7 | 0 | 10.3
  Pain Score: Severe | 2.9 | 0 | 1.5
  Healing Score: HemCon Better than Control | 0 | 0 | 14.7
  Healing Score: HemCon Same as Control | 0 | 0 | 29.4
  Healing Score: HemCon Worse than Control | 0 | 0 | 4.4
  Gingival Inflammation: None | 85.3 | 77.8 | 73.5
  Gingival Inflammation: Mild | 11.8 | 5.6 | 16.2
  Gingival Inflammation: Moderate | 0 | 11.1 | 7.4
  Gingival Inflammation: Severe | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for over the time in which the patient was in the care of the oral surgeon or was enrolled in the study. In most cases, the time frame for the subject was seven days.
Arm/Group | Hemcon Dental Dressing and Gauze With Pressure
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 20/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemcon Dental Dressing and Gauze With Pressure (N=71)
Dry Socket (General disorders) | 19 (19)
Packed Food (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No